CLINICAL TRIAL: NCT05662163
Title: Effect of General Anesthesia Method Chosen in Non-cardiac Surgery of Cardiac Risk Patients on Ischemia Modified Albumin and Heart-Type Fatty Acid-Binding Protein (H-FABP) Levels
Brief Title: Effect of General Anesthesia Method on Cardiac Risk Patients on Ischemia Modified Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: B.30.2.ATA.0.01.00/296
Record Dates: First submitted 2022-09-06; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP TIVA (Active Comparator): Anesthesia will be maintained with propofol (6-10 mg/kg/hour) and remifentanil (0.1-0.3 μg/kg/min). Blood will be taken from the patients at 0, 1 and 4 hours, centrifuged and stored at -80 degrees. From these examples, CK, CKMB, HIGH SENSITIVE TROPONIN, HFABP, IMA AND ALBUMIN will be studied.
  Interventions: Procedure: TIVA
- GROUP INHALATION ANESTHESIA (Active Comparator): Anesthesia will be maintained with sevoflurane (2 ml/min) 50% oxygen and remifentanil (0.1-0.3 μg/kg/min). Blood will be taken from the patients at 0, 1 and 4 hours, centrifuged and stored at -80 degrees. From these examples, CK, CKMB, HIGH SENSITIVE TROPONIN, HFABP, IMA AND ALBUMIN will be studied.
  Interventions: Procedure: GENERAL ANESTHESIA

INTERVENTIONS:
Procedure: TIVA — Anesthesia will be maintained with propofol (6-10 mg/kg/hour) and remifentanil (0.1-0.3 μg/kg/min).
  Arms: GROUP TIVA
Procedure: GENERAL ANESTHESIA — Anesthesia will be maintained with sevoflurane (2 ml/min) 50% oxygen and remifentanil (0.1-0.3 μg/kg/min).
  Arms: GROUP INHALATION ANESTHESIA

SUMMARY:
To examine the effects of the general anesthesia method chosen in non-cardiac surgical operations of patients with cardiac risk on the levels of cardiac markers

DETAILED DESCRIPTION:
To examine the effects of the general anesthesia method chosen in non-cardiac surgical operations of patients with cardiac risk on the levels of cardiac markers like; serum levels of the Creatine Kinase, Creatine Kinase Myocardial Band, high sensitive troponin, heart-type fatty acid-binding protein, ischemia-modified albumin and albumin. And evaluate the effect of anesthesia method on haemodynamic.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Getting a score of 2 and above according to the Lee cardiac index
* Having a non-cardiac surgical procedure that will take at least three hours
* ASA II or III

Exclusion Criteria:

* Under 18 years old
* Those who refused to participate in the study
* Patients with chronic renal failure
* Patients with creatinine value ≥ 1.5 mg/dl
* Surgery that takes less than 3 hours
* Patients with liver failure
* Refusing to participate in the study
* Being allergic to the drugs used

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
comparing serum levels of ischemia modified albumin | intraoperative period
  serum levels of ischemia modified albumin (in terms of IU/ML)
comparing serum levels of heart fatty acid binding protein | intraoperative period
  serum levels of heart fatty acid binding protein (in terms of mcg/L)

SECONDARY OUTCOMES:
The effect of anesthesia method used in cardiac risk patients in terms of ephedrine consumption | intraoperative period
  used ephedrine amount (mg)

CONTACTS AND LOCATIONS:
Overall Officials: Canan Atalat, Study Director — Ataturk University